CLINICAL TRIAL: NCT02145975
Title: Efficacy of Fentanyl to Reduce the Time of Severe Postoperative Pain Relief Compared to Morphine: a Randomized Parallel-group, Double-blind Clinical Trial
Brief Title: Efficacy of Fentanyl to Reduce the Time of Severe Postoperative Pain Relief Compared to Morphine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Olga Lucia Giraldo Salazar, MD, MSc, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDEAFEN001
Record Dates: First submitted 2014-05-18; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Postoperative Pain
Keywords: Severe postoperative pain; Morphine; Fentanyl; Time to titration of pain; Pain and PACU; Anesthesiology
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Fentanyl; Analgesics, Opioid; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl (Experimental): Procedure: Fentanyl for rescue of acute postoperative pain in the postanesthesia care unit
  Intervention:
  The nurse will administer 1 ug per kg during 5 seconds when the patient complain of pain (visual analog scale, VAS, ≥7). Immediately with the onset of drug administration a timer started; every 5 minutes the researcher assess the EVA and the drug will be administered if VAS > 3, until the patient manifests as a lower pain VAS ≤ 3 (mild). The nurse in charge in the PACU will manage the drug and will take 100 ug of fentanyl which is diluted in 10 mL of normal saline leaving a 10μg per ml concentration, are not labeled and for the physical and chemical characteristics of both drugs (colorless) risks of unblinded is minimized.
  Interventions: Drug: Fentanyl
- Morphine (Active Comparator): Procedure: Morphine for rescue of acute postoperative pain in the postanesthesia care unit
  Intervention:
  The nurse will administer 0,1 mg per kg during 5 seconds when the patient complain of pain (visual analog scale, VAS, ≥7). Immediately with the onset of drug administration a timer started; every 5 minutes the researcher assess the EVA and the drug will be administered if VAS > 3, until the patient manifests as a lower pain VAS ≤ 3 (mild). The nurse in charge in the PACU will manage the drug and will take 10 mg of morphine which is diluted in 10 mL of normal saline leaving a 1 mg per ml concentration, are not labeled and for the physical and chemical characteristics of both drugs (colorless) risks of unblinded is minimized.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Fentanyl — The nurse will administer 1 ug per kg during 5 seconds when the patient complain of pain (visual analog scale, VAS, ≥7). Immediately with the onset of drug administration a timer started; every 5 minutes the researcher assess the EVA and the drug will be administered if VAS > 3, until the patient manifests as a lower pain VAS ≤ 3 (mild). The nurse in charge in the PACU will manage the drug and will take 100 ug of fentanyl which is diluted in 10 mL of normal saline leaving a 10μg per ml concentration, are not labeled and for the physical and chemical characteristics of both drugs (colorless) risks of unblinded is minimized.
  Other Names: Opioids
  Arms: Fentanyl
Drug: Morphine — The nurse will administer 0,1 mg per kg during 5 seconds when the patient complain of pain (visual analog scale, VAS, ≥7). Immediately with the onset of drug administration a timer started; every 5 minutes the researcher assess the EVA and the drug will be administered if VAS > 3, until the patient manifests as a lower pain VAS ≤ 3 (mild). The nurse in charge in the PACU will manage the drug and will take 10 mg of morphine which is diluted in 10 mL of normal saline leaving a 1 mg per ml concentration, are not labeled and for the physical and chemical characteristics of both drugs (colorless) risks of unblinded is minimized.
  Other Names: Opioids
  Arms: Morphine

SUMMARY:
Fentanyl is a potent opioid, it is theoretically 100 times more potent that morphine and in severe acute postoperative pain acts faster than its congener (morphine ) for pain relief . In the literature there is no study that corroborates this theoretical assumption and proposes to compare which has fewer adverse effects. This drug produces effects similar to those reported for morphine but less magnitude and has the advantage that during the postoperative period respiratory depression, antitussive effect , gastrointestinal discomfort and physical dependence are manifested in a significantly less degree.

Trying to solve the management of postoperative pain relief , our objective is to determine by controlled clinical trial of superiority if in adult patients undergoing surgery , fentanyl reduces faster qualification time of severe pain to mild pain in the postanesthesia care unit compared to morphine.

DETAILED DESCRIPTION:
Postoperative pain is a severe problem of high incidence worldwide. According to a systematic review of the literature by Dolin et al , the incidence of moderate to severe postoperative pain in 41% of patients were found , and of these , only 23% experienced relief of the same ( 1). International Association for Study of Pain defines pain as unpleasant sensory or emotional experience associated with actual or potential damage , or described in terms of such damage ( 3). The postoperative pain is not only important for to cause suffering or unpleasant experience to the patient, but also by involving harmful effects to the body ( 4). Thus, the secondary stress to pain triggers the release of a series of hormonal mediators and activation of the sympathetic nervous system in conjunction with surgical trauma and previous comorbidities of the patient, that cause dysfunction of multiple organ systems , including the cardiovascular (5, 6) , GI (7-10) and respiratory ( 11,12 ), among others , increasing the incidence of postoperative complications such as myocardial ischemia , atelectasis ( 25-75 % after abdominal surgery) , respiratory infections (pneumonia 1-3 % after cardiac surgery ) , ileus , deep vein thrombosis and cognitive dysfunction. Thus increases the morbidity and patient recovery is delayed. (5) Similarly it has been observed that postoperative pain increases stay in the post anesthesia care unit , readmission for pain management, and delayed rehabilitation and reintegration of patients to activities of daily living , with the consequent increase in costs (5) . Considering the above arguments , it is obvious that timely intervention generates profit problem on multiple levels.

While the management of postoperative pain should include issues ranging from education to the patient prior to its analgesic plan to late recovery period in the post-anesthesia care area is crucial. This is because it has been shown that poor control of postoperative pain ( 3) in the early hours is associated with higher levels of pain at 48 hours . There is growing interest in the question of why , despite the availability of different drugs and technological advances that allow a better understanding of the pathophysiology of pain , has not been achieved a greater impact on the incidence of this problem ( 13).

Opioids are the most important drugs for postoperative pain control. In the post-anesthesia care area , especially when faced with a patient with severe or unbearable pain (14,15) , the analgesic opioid titration is the most effective strategy for controlling postoperative pain ( 16). The most studied and used today opioid is morphine, which by its pharmacokinetic characteristics provides an important balance between speed of onset and maintenance of analgesia ( 17). However, there are other alternatives for analgesic titration , such as fentanyl , which has favorable pharmacokinetics to have a faster response and thus may shorten the time needed to decrease pain from severe to mild ( 14,15). There are comparative studies between fixed-dose fentanyl and morphine in the emergency services and some preliminary tests in the recovery area (18,19). The most recent of analgesic titration trials comparing appropriate doses of opioids to patient weight which would improve its efficacy and safety ( 20). The tests that are known to have used fentanyl and morphine compared fixed-dose and 10 minute intervals .

Fentanyl is a potent opioid, it is theoretically 100 times more potent that morphine and in severe acute postoperative pain acts faster than its congener (morphine ) for pain relief . In the literature there is no study that corroborates this theoretical assumption and proposes to compare which has fewer adverse effects. This drug produces effects similar to those reported for morphine but less magnitude and has the advantage that during the postoperative period respiratory depression, antitussive effect , gastrointestinal discomfort and physical dependence are manifested in a significantly less degree.

Trying to solve the management of postoperative pain relief , our objective is to determine by controlled clinical trial of superiority if in adult patients undergoing surgery , fentanyl reduces faster qualification time of severe pain to mild pain in the postanesthesia care unit compared to morphine.

ELIGIBILITY:
Inclusion Criteria:

* Patients physical status I and IV, 18-65 years of age
* Patients scheduled for surgery under general or regional anesthesia and fasting as defined in the fasting guidelines.
* Patients whose accept and sign the informed consent of study.

Exclusion Criteria:

* Patients with severe respiratory depression given by a monitoring state indicating hypoxemia (oxyhemoglobin saturation below 90 %).

Patients with immediate postoperative hemodynamic instability given by bradycardia , hypotension or hypoperfusion states observed by clinical paleness, active bleeding, altered sensorium, and altered alertness not explained by effects of anesthetics .

Neurological disorders such as metabolic basis psychiatric disorders, mental retardation, congenital neurodegenerative conditions, hypoxic or ischemic related to aging that do not allow adequate evaluation of the analog scale pain assessment.

Patients with a history of tolerance to opioids for chronic use, which is defined to a period of 2 weeks.

Patients who have undergone epidural analgesia protocols, neuraxial and peripheral nerve blocks.

Patients with any alteration in neurological status. History of psychiatric disorders. Patient with known hypersensitivity or allergic reactions to opioids. Women who are pregnant or suspected to be.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Time in minutes of titration of fentanyl and morphine in reducing severe postoperative pain to mild pain | The outcome will be measured from the patient presents severe pain at the PACU until the time that presents mild pain and he does not need more rescue bolus assessed up to 4 hours
  Time in minutes of titration of fentanyl and morphine in reducing postoperative pain severe to mild pain with visual analog scale (≤ 3).

SECONDARY OUTCOMES:
Stay time of patients in the postanesthetic recovery unit in hours. | The outcomes will be measured from the patient arrives at the PACU until he is discharged or transferred to the hospital room assessed up to 4 hours.
  Stay time of patients in the postanesthetic recovery unit in hours.
Satisfaction with the analgesic management | This outcome will be measured in the first hour at the PACU and postoperative 24 hours
  Satisfaction with the analgesic management received by the Likert scale in both groups at the time and 24 hours.
Cumulative dosis | The outcome will be measured from the patient experiences severe pain at the PACU and is given the first bolus rescue analgesic until is given last bolus rescue analgesic, assessed up to 4 hours
  Cumulative dose of fentanyl vs morphine required for relief of pain in both groups.
Saturation of oxygen and arterial pressure | The outcomes will be measured from the patient arrives at the PACU until he is discharged or transferred to the hospital room, assessed up to 4 hours.
  O2 saturation and MAP in both groups every 5 minutes during the titration period.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Cadavid, MD, Principal Investigator — Antioquia University
Locations (1):
- Antioquia University, Medellín, Antioquia, Colombia